CLINICAL TRIAL: NCT01042080
Title: Effect of Mechanical Ventilation With NAVA and PSV on Inspiratory Muscle Workload and Synchrony in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Neurally Adjusted Ventilatory Assist and Synchrony in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: NAVASYNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Principal Investigator, Jerome Allardet-Servent, MD, MD, MSc, Hôpital Européen Marseille
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2009-A01099-48
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Mechanical ventilation; Neurally adjusted ventilatory assist (NAVA); Acute respiratory failure; Chronic obstructive pulmonary disease; Weaning; Invasive mechanical ventilation; Positive Pressure support Ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PSV-ET 25 (Active Comparator): Pressure support ventilation with expiratory trigger set at 25 %.
  Interventions: Other: Expiratory trigger (ET)
- PSV-ET 50 (Active Comparator): Pressure support ventilation with expiratory cycling set at 50 %.
  Interventions: Other: Expiratory trigger (ET)
- NAVA (Experimental): NAVA level is adjusted to achieve similar peak inspiratory pressure levels than during PSV.
  Interventions: Device: NAVA

INTERVENTIONS:
Device: NAVA — Assisted mechanical ventilation according to the electrical activity of the diaphragm recorded with a 16-FR naso-gastric tube mounted with EMG electrodes
  Other Names: Neurally Adjusted Ventilatory Assist
  Arms: NAVA
Other: Expiratory trigger (ET) — Varying the cycling criterion according to the percentage of peak inspiratory flow
  Arms: PSV-ET 25; PSV-ET 50

SUMMARY:
NAVA used the electrical activity of the diaphragm (EAdi) to initiate and deliver in proportion of an inspiratory assistance. During inspiration, EAdi signal occurred earlier than airflow or pressure variations in the airway. The investigators hypothesized that NAVA improved patient-ventilator synchrony and reduced inspiratory workload as compared with pressure support ventilation delivered at two different cycling criteria (25 and 50 %).

ELIGIBILITY:
Inclusion Criteria:

* History of chronic obstructive pulmonary disease
* Admitted for acute respiratory failure requiring invasive mechanical ventilation
* Currently receiving pressure support ventilation

Exclusion Criteria:

* Age < 18 years
* Respiratory rate > 35 bpm
* Severe hypoxemia with SpO2 < 88 % and FIO2 > 50 %
* Heart rate > 120 bpm
* Systolic arterial pressure < 90 mmHg
* Contraindication to naso-gastric tube's insertion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Inspiratory muscle workload as reflected by the diaphragmatic Pressure Time Product (PTPdi) | 5 minutes

SECONDARY OUTCOMES:
Ineffective inspiratory effort | 5 minutes
Dynamic intrinsic PEEP | 5 minutes
Arterial blood gases | 20 minutes
Trigger delay | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme ALLARDET-SERVENT, MD, MSc, Principal Investigator — Fondation Hôpital Ambroise Paré
Locations (2):
- France (2):
  - Hopital Paul Desbief, Marseille
  - Fondation Hôpital Ambroise Paré, Marseille